CLINICAL TRIAL: NCT06974591
Title: Postural Perturbations Tracing to the Stomatognathic System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H-45251
Record Dates: First submitted 2025-05-08; First posted 2025-05-16 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Posture
Keywords: Dental splints; Dentures; Vertical Dimension of Occlusion; Temporomandibular Joint Disorders; Balance; Gait
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Occlusal Splints; Dentures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A- dental splints (Active Comparator): Participants in this group will be adults aged 30-45 with complete dentition and Class I malocclusion. Participants must have a complete set of teeth, either natural or with crowns, ensuring no teeth are missing.
  Interventions: Other: Dental splints
- Group B- dentures (Active Comparator): Participants in this group will be older adults aged 50-65 who are edentulous (without natural teeth) and wear full dentures.
  Interventions: Other: Dentures

INTERVENTIONS:
Other: Dental splints — Each participant will receive six custom-made dental splints to incrementally increase their VDO. These splints will alter the VDO in increments from 5 to 30 mm, specifically: 5, 10, 15, 20, 25, and 30 mm.
  Arms: Group A- dental splints
Other: Dentures — Participants in this group will participate in balance and gait testing both with and without their dentures to examine how the presence or absence of dentures affects postural stability and movement.
  Arms: Group B- dentures

SUMMARY:
A connection of the stomatognathic system [an anatomical system comprising the teeth, jaws, and associated soft tissues] to postural control has been suggested in the literature. This research will investigate how occlusion can impact postural response, disorder, and rehabilitation by examining how modifications in the vertical dimension of occlusion (VDO) influence balance and gait.

Although it is currently unclear which or how restorative approaches cause postural disturbances, changes in several occlusal factors, i.e. VDO, Angle's class, crossbite and others have been suggested to manifest clearly into an altered stability, which could have a significant effect on the quality of life, especially in the elderly.

The present study aims to identify the degree to which specific interventions in oral cavity affect the stability and gait patterns of patients, This will b achieved by either:

* The use of dental splints (fully certified devices)
* The use of the subjects' own dentures

A direct correlation of postural perturbations and VDO, would essentially void the necessity to evaluate specific interventions (e.g. different types of restorations) independently and allow clinicians to assess a potential effect on their patients' stability and gait based on pre- to post- treatment VDO.

ELIGIBILITY:
Inclusion Criteria for Group A

* 30-45 years old
* Physically and cognitively healthy (able to easily walk without assistance)
* Possessing a complete set of teeth (either natural or restored with crowns)
* Classified as Class I malocclusion according to Angle's criteria.

Inclusion criteria for Group B

* 50-65 years old
* Physically and cognitively healthy (able to easily walk without assistance)
* Fully edentulous
* Wear complete dentures

Exclusion Criteria:

* Parkinson's Disease
* Morbid obesity i.e. BMI values exceeding 40, calculated based on body weight and height requested over the phone or during the visit
* Occlusion altered due to a non-physiological condition i.e. trauma or pathology
* Active temporomandibular joint disorder
* Pregnancy, as pregnancy-related physiological changes could influence the study's balance and gait measurements. This exclusion will be based on self-report during the screening process, and no additional testing will be conducted.
* Any other condition that in the opinion of the study researchers has potential to impact balance or gait

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Center of pressure | 60-90 minutes
  This outcome will be assessed from data collected with a motion capture system (consisting of specialized infrared cameras), which will document the kinematics of reflective markers, placed on the subjects' head and body.
Postural sway | 60-90 minutes
  This outcome will be assessed from data collected with a motion capture system (consisting of specialized infrared cameras), which will document the kinematics of reflective markers, placed on the subjects' head and body.
Stride length | 60-90 minutes
  This outcome will be assessed from data collected with a motion capture system (consisting of specialized infrared cameras), which will document the kinematics of reflective markers, placed on the subjects' head and body.
Step width | 60-90 minutes
  This outcome will be assessed from data collected with a motion capture system (consisting of specialized infrared cameras), which will document the kinematics of reflective markers, placed on the subjects' head and body.
Gait velocity | 60-90 minutes
  This outcome will be assessed from data collected with a motion capture system (consisting of specialized infrared cameras), which will document the kinematics of reflective markers, placed on the subjects' head and body.
Muscle activation | 60-90 minutes
  This outcome will be assessed from data collected with wireless Electromyography (consisting of small sensors), which will document the activation of specific muscle groups, controlling head and jaw position.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Tsouknidas, PhD, Principal Investigator — Goldman School of Dental Medicine, Boston University
Locations (1):
- Goldman School of Dental Medicine, Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No